CLINICAL TRIAL: NCT06299826
Title: A Phase IIb Two-Cohort, Randomised, Placebo-controlled, Double-blind, Multi-centre, Dose-ranging Study of AZD5462 in Stable Patients With Chronic Heart Failure
Brief Title: A Phase IIb Study of AZD5462 in Patients With Chronic Heart Failure
Acronym: LUMINARA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9090C00008; 2023-510148-19-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-02-16; First posted 2024-03-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Chronic Heart Failure
Keywords: Relaxin Family Peptide Receptor 1 (RXFP1) agonist

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A & B: AZD5462 low dose (Experimental): Participants will receive low dose of AZD5462 as OD tablets for 24 weeks.
  Interventions: Drug: AZD5462
- Cohort A & B: AZD5462 medium dose (Experimental): Participants will receive medium dose of AZD5462 as OD tablets for 24 weeks.
  Interventions: Drug: AZD5462
- Cohort A & B: AZD5462 high dose (Experimental): Participants will receive high dose of AZD5462 as OD tablets for 24 weeks.
  Interventions: Drug: AZD5462
- Cohort A & B: Placebo (Experimental): Participants will receive matching placebo OD tablets for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5462 — Participants will receive low, medium & high doses of film-coated tablets of AZD5462 OD orally.
  Arms: Cohort A & B: AZD5462 high dose; Cohort A & B: AZD5462 low dose; Cohort A & B: AZD5462 medium dose
Drug: Placebo — Participants will receive matching doses of film-coated tablets of Placebo OD orally.
  Arms: Cohort A & B: Placebo

SUMMARY:
The main purpose of this study is to evaluate the effect of AZD5462 on cardiac function in participants with chronic heart failure (HF).

DETAILED DESCRIPTION:
This is a Phase IIb randomized, double-blind, placebo-controlled, multi-center, dose-ranging study to evaluate the efficacy, safety, and pharmacokinetic (PK) of AZD5462 on top of standard of care in 2 cohorts of participants with HF: Cohort A, and Cohort B.

The study will include 3 periods and approximately 12 study visits:

* Screening period of up to 4 weeks (at least 1 study visit)
* Treatment period of 24 weeks (8 study visits)
* Follow-up period of 4 weeks (3 study visits)

Eligible participants in each cohort will be randomized equally 1:1:1:1 to receive a once daily dose (OD) of 3 dose levels (low, medium, or high) oral dose of AZD5462 tablets or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a pre-existing diagnosis of HF NYHA FC II to IV.
* Participants must be on stable HF standard of care medication for at least 4 weeks prior to consent and during the Screening period.
* Minimum body mass index (BMI) of 18 kilograms per meter square (kg/m^2) at Screening.
* For female participants, the participant must not be pregnant or lactating and must be of non-childbearing potential.
* All male participants should refrain from fathering a child or donating sperm until 3 months after the final study Follow-up Visit. Non-sterilised male participants should avoid fathering a child either by true abstinence or use of a condom for all sexual intercourse with a female partner of childbearing potential from the first dose until 3 months after the final Follow-up Visit.

Exclusion Criteria:

* Historical or current evidence of a clinically significant disease or disorder including, but not limited to:

  1. Myocardial infarction, stroke, transient ischaemic attack, coronary artery bypass grafting, or percutaneous coronary intervention within 12 weeks prior to consent or transcatheter structural heart interventions or cardiac valve surgery within 6 months prior to consent.
  2. Sarcoidosis, restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, or hypertrophic (obstructive) cardiomyopathy.
  3. History of untreated clinically significant valve disease or a Screening confirmation of severe aortic stenosis, severe mitral stenosis, moderate or severe aortic insufficiency or severe mitral insufficiency.
  4. Amyloidosis, Fabry disease, or haemochromatosis.
  5. Pericardial disease (i.e., visually significant white pericardium on echocardiogram).
  6. Known coagulation disorders.
  7. Current diagnosis of active hepatitis.
  8. Severe pulmonary disease that is not expected to improve over time, as assessed by the investigator.
  9. Decompensated HF or any cardiopulmonary hospitalisation, except planned hospitalisation without worsening of cardiac or pulmonary functions, within 4 weeks prior to consent or during the Screening period.
  10. History of active malignancy within 2 years, except for fully excised or treated basal cell carcinoma, or ≤ 2 squamous cell carcinomas of the skin and participants who are under investigation for breast or cervical cancer, including participants with a pap smear of grade ≥ 3.
* History of hypersensitivity to AZD5462 or any component of AZD5462 drug product.
* Known history of drug or alcohol abuse within 24 months of Screening.
* Congenital long QT syndrome or history of QT prolongation associated with other medications that required discontinuation of that medication.
* Cardiac ventricular arrhythmia that requires treatment.
* History of or anticipated heart transplant.
* Current or planned cardiac resynchronization therapy/bi-ventricular pacemaker or mechanical assist device implantation.
* Any planned highly invasive cardiovascular procedure (eg, coronary revascularisation, ablation of atrial fibrillation/flutter etc).
* Positive hepatitis C antibody, or hepatitis B virus surface antigen at Screening. Participants with positive hepatitis B virus core antibody can be included in the study as long as hepatitis B virus surface antigen is negative, and there are no other signs of an active hepatitis B.
* Known to have historically tested positive for Human Immunodeficiency Virus.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Cohort A and B: Change from Baseline in Echocardiography Parameters | From Baseline to Week 25
  To evaluate the effect of AZD5462 after treatment in participants with HF.

SECONDARY OUTCOMES:
Cohort A and B: Change from Baseline in Echocardiography Parameters | From Baseline to Week 13 and Week 25
  To evaluate the effect and dose response of AZD5462 and effect on echocardiographic markers related to structural, systolic and diastolic function after treatment in participants with HF.
Cohorts A and B: Change from Baseline in Kansas City Cardiomyopathy Questionnaire overall summary score (KCCQ-OSS) | From Baseline to Weeks 3, 5, 13, and 25
  To evaluate the effect of AZD5462 on HF health status in participants with HF.
  The KCCQ is a validated questionnaire developed for patients with congestive HF. It is a 23-item, self-administered health status measure that quantifies physical limitations, symptoms, social interference, self-efficacy, and quality of life. Results for each domain are summarized and transformed to a score of 0 to 100 with higher scores indicating better health status.
Cohorts A and B: Change from Baseline in New York Heart Association Functional Class (NYHA FC) | Baseline and Week 25
  To evaluate the effect of AZD5462 on HF health status in participants with HF.
  The NYHA Functional Classification is a system to measure the severity of symptoms of heart failure. It places patients in four categories based on limitations of physical activity, from Class I with no limitation, progressing to Class IV with severe limitations.
Cohorts A and B: Change from Baseline in cardiac biomarkers | From Baseline to Weeks 5, 13, and 25
  To evaluate the effect of AZD5462 on biomarkers of cardiac function in treatment participants with HF.
Cohorts A and B : Plasma Concentration of AZD5462 | Day 15 (Week 3), Day 29 (Week 5) and 85 (Week 13)
  To evaluate the PK of AZD5462 after repeat OD oral dosing in participants with HF.
Cohorts A and B: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Baseline to Week 29 (Day 197)
  To evaluate the safety and tolerability of AZD5462 as compared to placebo in participants with HF.

CONTACTS AND LOCATIONS:
Locations (51):
- United States (14):
  - Research Site, Alexander City, Alabama
  - Research Site, Northridge, California
  - Research Site, Torrance, California
  - Research Site, Vista, California
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Richmond, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Buffalo, New York
  - Research Site, Rosedale, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Manassas, Virginia
- Bulgaria (2):
  - Research Site, Pleven
  - Research Site, Sofia
- Czechia (5):
  - Research Site, Brno
  - Research Site, Jaroměř
  - Research Site, Liberec
  - Research Site, Louny
  - Research Site, Pilsen
- Denmark (2):
  - Research Site, Aalborg
  - Research Site, Herning
- Hungary (4):
  - Research Site, Balatonfüred
  - Research Site, Kistarcsa
  - Research Site, Nyíregyháza
  - Research Site, Székesfehérvár
- India (4):
  - Research Site, Kochi
  - Research Site, Kolkata
  - Research Site, Surat
  - Research Site, Vadodara
- Japan (11):
  - Research Site, Fukui-shi
  - Research Site, Higashiibaraki-gun
  - Research Site, Higashiohmi-shi
  - Research Site, Kitakyushu
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Miyazaki
  - Research Site, Morioka
  - Research Site, Naha
  - Research Site, Ōmihachiman
  - Research Site, Shūnan
- Netherlands (3):
  - Research Site, Breda
  - Research Site, Deventer
  - Research Site, Enschede
- Poland (4):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Košice

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/